CLINICAL TRIAL: NCT01603329
Title: Increasing Medication Adherence Through Physician Incentives and Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Humana Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 007
Record Dates: First submitted 2012-05-16; First posted 2012-05-22 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Medication Adherence
Keywords: medication adherence; diabetes; hypertension; cholesterol; statins
MeSH Terms: conditions — Medication Adherence; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Comprehensive incentives + comprehensive communication (Experimental): Physicians are given financial incentives for improving patient medication adherence for all of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, and cholesterol (statins) medication.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Comp incentives + comp communication + non-white paper (Experimental): Physicians are given financial incentives for improving patient medication adherence for all of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, and cholesterol (statins) medication, and their patient reports are printed on non-white bright colored paper.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Focused incentives + focused com for oral diabetes medication (Experimental): Physicians are given financial incentives for improving patient medication adherence for oral diabetes medication.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Foc incentives + foc comm for Diabetes + non-white paper (Experimental): Physicians given financial incentives for improving patient medication adherence for oral diabetes medication and patient reports are printed on bright non-white paper.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Focused incentives + focused comm for hypertension meds (Experimental): Physicians are given financial incentives for improving patient medication adherence for hypertension (ACEI or ARB) medication.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Foc incentives + comm for hypertension meds + non-white paper (Experimental): Physicians are given financial incentives for improving patient medication adherence for hypertension (ACEI or ARB) medication with patient reports on non-white paper.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Focused incentives + focused comm for cholesterol meds (Experimental): Physicians given financial incentives for improving patient medication adherence for cholesterol (statins) medication.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Foc incentives +comm for cholesterol meds + non-white paper (Experimental): Physicians given financial incentives for improving patient medication adherence for cholesterol (statins) medication and patient reports are printed on non-white paper.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Comprehensive communiation (Experimental): Physicians are given communication emphasizing the importance of improving adherence to all of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, and cholesterol (statins) medication.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Comprehensive communication + non-white paper (Experimental): Physicians are given communication emphasizing the importance of improving adherence to all of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, and cholesterol (statins) medication and patient reports are printed on non-white paper.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging
- Control Arm (Experimental): Physicians and their patient adherence is tracked, but they receive no intervention.
  Interventions: Other: Increasing Medication Adherence through Physician Incentives and Messaging

INTERVENTIONS:
Other: Increasing Medication Adherence through Physician Incentives and Messaging — There are two treatments:
  1. Physicians given financial incentives for improving patient medication adherence for all of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, and cholesterol (statins) medication vs. one of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, or cholesterol (statins) medication.
  2. Physicians given communication emphasizing the importance of improving adherence to all of the previous medication classes vs. one one of the previous medication classes.
  When physicians are sent a communication regarding the opportunity to receive an incentive as part of our pilot, they will also receive a single patient sheet for each patient who has less than 80% adherence. For half of the arms, the investigators will make the patient sheets a bright, non-white, color, in order to further draw the physicians' attention to that specific paper in their chart.
  Other Names: Adherence

SUMMARY:
The goal of this project is to increase patient adherence to medication using communications and incentives for physicians. The investigators are partnering with a health insurance company, Humana Inc, to design and implement an incentives program for physicians whose patients increase their medication adherence for oral diabetes medication, hypertension (ACEI or ARB) medication, and/or cholesterol (statins) medication. The investigators will use behavioral economics to explore the best way to communicate the incentives to the physicians.

DETAILED DESCRIPTION:
Traditional economics would suggest that the best way to maximize adherence would be to give physicians financial incentives to improve adherence to all relevant drugs, and that communications to physicians should emphasize all of the relevant drugs. Behavioral economics suggests theory suggests that if you emphasize everything, then you are effectively emphasizing nothing. Behavioral econonmics would suggest to maximize adherence one should give physicians financial incentives for improving adherence for a small number of relevant drugs, and communications to physicians should emphasize a small number of the relevant drugs. This allows physicians to focus their energy and reduces the probability that they will give up because they're overwhelmed, or in other words, avoid the phenomenon called metric fatigue.

Humana has already implemented an incentives program for physicians, and the investigators will work with them to design a program that just focuses on medication adherence. Physicians targeted for this pilot could also be enrolled in another Humana incentives program, but this incentives program will act independently of the other.

There are two treatment dimensions the investigators will test via random assignment at the practice level:

1. Physicians given financial incentives for improving patient medication adherence for all of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, and cholesterol (statins) medication vs. one of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, or cholesterol (statins) medication.
2. Physicians given communication emphasizing the importance of improving adherence to all of the previous medication classes vs. one one of the previous medication classes.

In a previous study to increase uptake of colonoscopies among employees at a partner firm, the investigators found that using a post it note to catch the attention of the employee statistically significantly increased colonoscopy uptake over a control group. The investigators will also employ an eye catching method in the proposed pilot. When physicians are sent a communication regarding the opportunity to receive an incentive as part of our pilot, they will also receive a single patient sheet for each patient who has less than 80% adherence. They will be encouraged to include the patient sheet in their chart as a reminder to discuss medication adherence with their patient the next time they see them. For half of our arms, the investigators will make the patient sheets a bright, non-white, color, in order to futher draw the physicians' attention to that specific paper in their chart.

Our experimental arms will be:

1. Comprehensive incentives + comprehensive communication
2. Comprehensive incentives + comprehensive communication + printed on bright non-white paper
3. Focused incentives + focused communication (one for all three drug classes)
4. Focused incentives + focused communication + printed on bright non-white paper (one for all three drug classes)
5. Comprehensive communiation
6. Comprehensive communication + printed on bright non-white paper
7. Control arm: no communication + no incentives

The investigators hypothesize that physicians who receive focused incentives and focused communications will have more patients with increased medication adherence than physicians who receive comprehensive incentives and comprehensive communications. The investigators also hypothsize that physicians who receive patient sheets using bright, non-white paper will have more patients with increased medication adherence than physicians who receive plain white patient sheets.

ELIGIBILITY:
Inclusion Criteria:

* Physician in the Humana network
* Treats Humana Medicare Advantage Members
* Has Humana Medicare Advantage members who are taking at least one of the following medications: oral diabetes medication, hypertension (ACEI or ARB) medication, and/or cholesterol (statins) medication, and who are less than 80% adherent.

Exclusion Criteria:

* Practices with more than 10 physicians

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 734 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | Up to two years
  The investigators will see how the treatment arms affect the targeted physicians' patients medication adherence for oral diabetes medication, hypertension (ACEI or ARB) medication, and cholesterol (statins) medication.

SECONDARY OUTCOMES:
Demographic Controls for Physicians | Up to two years
  The investigators will see if our targeted physicians' demographic controls affect their patients' medication adherence rates before and after treatment.
Demographic Controls for Patients | Up to 2 years
  The investigators will see how demographic controls for patients affect our targeted physicians' patients' medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: David I Laibson, Ph.D., Principal Investigator — National Bureau of Economic Research, Harvard University
Locations (1):
- Humana, Inc, Louisville, Kentucky, United States